CLINICAL TRIAL: NCT02277717
Title: A Two Part First-in-human Phase I Study (With Expanded Cohorts) With the Antibody-drug Conjugate SYD985 to Evaluate the Safety, Pharmacokinetics and Efficacy in Patients With Locally Advanced or Metastatic Solid Tumors
Brief Title: First-in-human Study With the Antibody-drug Conjugate SYD985 to Evaluate Safety and Efficacy in Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SYD985.001
Record Dates: First submitted 2014-10-21; First posted 2014-10-29 (Estimated); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Solid Tumors
Keywords: cancer; metastasis; HER2; trastuzumab; duocarmycin; SYD985; antibody-drug conjugate; ADC; trastuzumab vc-seco-DUBA
MeSH Terms: conditions — Neoplasms; Neoplasm Metastasis | interventions — trastuzumab duocarmazine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- SYD985 (trastuzumab vc-seco-DUBA) (Experimental): HER2-targeting Antibody-Drug Conjugate
  Interventions: Drug: SYD985 (trastuzumab vc-seco-DUBA)

INTERVENTIONS:
Drug: SYD985 (trastuzumab vc-seco-DUBA) — IV (in the vein) infusion every three weeks. Number of Cycles: until cancer progression or unacceptable toxicity develops. Different doses.

SUMMARY:
The purpose of this study is to evaluate the safety of a new medicinal drug SYD985 at different dose levels in patients with cancer, to understand how SYD985 is handled by the body and to evaluate the effect of SYD985 on the cancer.

DETAILED DESCRIPTION:
Cancer cells can have different kinds of proteins on their cell surface; one of these is the protein HER2. HER2 plays an important role in the development of cancer. High expression of HER2 is related to poor prognosis. Although several cancer drugs are available that work via the HER2 protein, a substantial portion of these patients still does not benefit from these treatments.

The new cancer drug SYD985 is being developed by Synthon Biopharmaceuticals B.V. SYD985 is an antibody-drug conjugate and consists of two parts: an antibody and a linker-drug moiety containing a toxin. The antibody part binds to HER2 on the surface of the cancer cell. When SYD985 binds to this cancer cell, it will be internalized by the cell. After proteolytic cleavage of the linker, the toxin will be split off in the cell and the cancer cell will be killed. Thus, SYD985 can be considered as a form of targeted chemotherapy.

This is the first study in which SYD985 is administered to humans. The study consists of two parts:

Part I is the dose-escalation part in which a low dose of SYD985 is given to three cancer patients. If it is well tolerated, a higher dose of SYD985 will be given to 3 other cancer patients. This will continue until a further dose increase is not safe anymore.

In Part II of the study, several groups of patients with a specific type of cancer will receive the SYD985 dose which has been selected for further evaluation.

All patients from both parts of the study will receive SYD985 infusions every three weeks until progression of the cancer or unacceptable toxicity develops.

ELIGIBILITY:
Main Inclusion Criteria:

1. Patient with histologically-confirmed, locally advanced or metastatic tumor who has progressed on standard therapy or for whom no standard therapy exists, with the following restriction:

   * Part I: solid tumors of any origin;
   * Part II: breast, gastric, urothelial and endometrial tumors;
2. For Part II: HER2 tumor status as defined in the protocol;
3. ECOG performance status ≤ 1;
4. Life expectancy > 12 weeks;
5. Adequate organ function;
6. For Part II: measurable disease.

Main Exclusion Criteria:

1. Anthracycline treatment within 3 months and/or abnormal cardiac biomarker values;
2. Other anticancer therapy (except for LHRH agonists) within 4 weeks (6 weeks for nitrosoureas and mitomycin C);
3. History of infusion-related reactions and/or hypersensitivity to trastuzumab or (ado-) trastuzumab emtansine;
4. Severe, uncontrolled systemic disease;
5. LVEF < 55%, or a history of absolute decrease in LVEF of ≥ 10% points to < 50% during previous treatment with trastuzumab or (ado-)trastuzumab emtansine, or a history of decrease in LVEF to < 40% during previous treatment with trastuzumab or (ado-)trastuzumab emtansine;
6. History of clinically significant CV disease;
7. Symptomatic brain metastasis, or therapy for brain metastasis (excluding PCI and dexamethasone treatment with stable or decreasing daily dose) within 4 weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 185 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2019-01 (Actual); Study Completion 2019-10 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | 21 days
  first cycle

SECONDARY OUTCOMES:
Number of patients with adverse events | up to 2 years
Area under the plasma concentration versus time curve (AUC) of SYD985 | Baseline, Days 1,2,3,4,8,15 of Cycle 1, Days 1,8,15 of Cycle 2, Day 1 of subsequent cycles up to 2 years
Peak plasma concentration of SYD985 | Baseline, Days 1,2,3,4,8,15 of Cycle 1, Days 1,8,15 of Cycle 2, Day 1 of subsequent cycles up to 2 years
Change from baseline in hematology and blood chemistry parameters | Baseline and every cycle up to 2 years
Number of patients with antibodies against SYD985 | Baseline and every cycle up to 2 years
Objective response rate | Baseline and every two cycles up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Mommers, PhD, Study Director — Synthon Biopharmaceuticals B.V., The Netherlands
Locations (15):
- Belgium (3):
  - UZ, Antwerp
  - Institut Jules Bordet, Brussels
  - UZ, Ghent
- Netherlands (4):
  - NKI-AvL, Amsterdam
  - UMC, Groningen
  - Radboud UMC, Nijmegen
  - UMC, Rotterdam
- Spain (4):
  - Institut Catala d'Oncologia, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - START Madrid-CIOCC, Madrid
  - START Madrid-FJD, Madrid
- United Kingdom (4):
  - Beatson Institute for Cancer Research, Glasgow
  - The Christie NHS Foundation Trust, Manchester
  - Churchill Hospital, Oxford
  - Royal Marsden / Institute of Cancer Research, Sutton

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Banerji U, van Herpen CML, Saura C, Thistlethwaite F, Lord S, Moreno V, Macpherson IR, Boni V, Rolfo C, de Vries EGE, Rottey S, Geenen J, Eskens F, Gil-Martin M, Mommers EC, Koper NP, Aftimos P. Trastuzumab duocarmazine in locally advanced and metastatic solid tumours and HER2-expressing breast cancer: a phase 1 dose-escalation and dose-expansion study. Lancet Oncol. 2019 Aug;20(8):1124-1135. doi: 10.1016/S1470-2045(19)30328-6. Epub 2019 Jun 27. PMID 31257177
- [Derived] Menderes G, Bonazzoli E, Bellone S, Black J, Altwerger G, Masserdotti A, Pettinella F, Zammataro L, Buza N, Hui P, Wong S, Litkouhi B, Ratner E, Silasi DA, Huang GS, Azodi M, Schwartz PE, Santin AD. SYD985, a novel duocarmycin-based HER2-targeting antibody-drug conjugate, shows promising antitumor activity in epithelial ovarian carcinoma with HER2/Neu expression. Gynecol Oncol. 2017 Jul;146(1):179-186. doi: 10.1016/j.ygyno.2017.04.023. Epub 2017 May 1. PMID 28473206